CLINICAL TRIAL: NCT06127992
Title: Photoplethysmography for Non-invasive Diagnosis of Cold Urticaria
Brief Title: Non-invasive Diagnosis of Cold Urticaria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: City Clinical Hospital No.52 of Moscow Healthcare Department (Other)
Responsible Party: Principal Investigator, Daria Fomina, Head of the Center of Allergy and Immunology, City Clinical Hospital No.52 of Moscow Healthcare Department
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06/0621
Record Dates: First submitted 2023-09-18; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Urticaria Cold
MeSH Terms: conditions — Cold Urticaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Typical ColdU (Experimental): 39 patients had typical ColdU confirmed by positive ICT and TempTest® CSTs.
  Interventions: Device: Cold stimulation tests / critical temperature threshold
- Atypical ColdU (Experimental): 24 patients had atypical ColdU with negative ICT and TempTest® CSTs.
  Interventions: Device: Cold stimulation tests / critical temperature threshold
- Control group (Other): 15 healthy controls (HCs) who had no history of pathological reactions associated with cold exposure, and all of them had negative CSTs
  Interventions: Device: Cold stimulation tests / critical temperature threshold

INTERVENTIONS:
Device: Cold stimulation tests / critical temperature threshold — ICT was performed following a standard protocol. Briefly, a melting ice cube in thin plastic bag was placed on the volar surface of the patient forearm for 5 min, with macroscopic assessment of the test site 10 min later. TempTest® CSTs were done with TempTest® 4.0 (Courage & Khazaka, Cologne, Germany), which has a single Peltier element (length: 350 mm, width: 2 mm) that provides a continuous temperature gradient from 4°C to 44°C. The use of TempTest® allows for reproducible and standardized cold (and heat) provocation tests and the identification of CTTs. TempTest® CST results were also assessed 10 min after the end of cold exposure.

SUMMARY:
The investigators subjected 63 patients (39 with typical Cold urticaria and 24 with atypical Cold urticaria ) and 15 healthy controls to TempTest® cold stimulation tests and critical temperature threshold assessments. Blood microcirculation photoplethysmography measurements were performed 5 min before and 10 min after the ice cube on the volar forearm.

ELIGIBILITY:
Inclusion Criteria:

* Cold urticaria

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-11-27 (Estimated); Study Completion 2023-11-27 (Estimated)

PRIMARY OUTCOMES:
Photoplethysmography amplitude | 10 min after the end of cold exposure
  To compute the blood flow signal, we subtracted slowly time-varying background and frequency components out of the cardiovascular-related range of 0.3-7 Hz. The resulting well-matched, noise-free and intensity-corrected blood flow images are suited for PPG calculation by averaging the intensity pixel values of each frame. The PPG amplitude is proportional to the amount of arterial blood that reaches the visualized skin area and thus characterizes its blood perfusion. It is measured in arbitrary units (AU). We performed photoplethysmographic assessments of the volar forearm of all patients 5 minutes before and 10 minutes after the beginning and end of ice cube application.

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow City Clinical Hospital 52, Moscow, Russia